CLINICAL TRIAL: NCT00014300
Title: Open Label Phase II Study On Glufosfamide Administered As A 60 Minute Infusion Every 3 Weeks In Recurrent Glioblastoma Multiforme
Brief Title: Glufosfamide in Treating Patients With Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-16994G-26002; EORTC-16994G-26002
Record Dates: First submitted 2001-04-10; First posted 2004-03-17 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Gliosarcoma | interventions — beta-D-glucosylisophosphoramide mustard

INTERVENTIONS:
Drug: glufosfamide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of glufosfamide in treating patients who have recurrent glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the activity of glufosfamide, in terms of objective response rate and/or progression-free survival at 6 months, in patients with recurrent glioblastoma multiforme. II. Determine the duration of objective response in patients treated with this regimen. III. Determine the toxic effects and pharmacokinetic profile of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients receive glufosfamide IV over 60 minutes on day 1. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients with stable disease receive treatment for a minimum of 6 months or until progression. Patients with an objective complete response receive a maximum of 2 additional courses of treatment after confirmation of response. Patients are followed every 6 weeks until progression.

PROJECTED ACCRUAL: A total of 28 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed glioblastoma multiforme Recurrent disease by CT scan or MRI At least 1 bidimensionally measurable target lesion at least 2 cm in the largest diameter

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: Neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 1.5 times upper limit of normal (ULN) Alkaline phosphatase no greater than 2.5 times ULN AST and ALT no greater than 2.5 times ULN Renal: Creatinine no greater than 1.5 mg/dL Creatinine clearance at least 60 mL/min Cardiovascular: Cardiac function normal No history of ischemic heart disease within the past 6 months 12 lead ECG normal Other: No other prior or concurrent malignancy except cone biopsied cervical cancer or adequately treated basal cell or squamous cell skin cancer No unstable systemic disease No active uncontrolled infection No psychological, familial, sociological, or geographical condition that would preclude study Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent prophylactic growth factors (e.g., filgrastim (G-CSF)) Chemotherapy: No more than 1 prior chemotherapy regimen as adjuvant therapy or for recurrent disease At least 6 weeks since prior chemotherapy Endocrine therapy: Stable or decreasing dose of corticosteroids for at least 1 week prior to study Radiotherapy: At least 3 months since prior radiotherapy to the brain No prior high-dose radiotherapy (more than 65 Gy), stereotactic radiosurgery, or internal radiotherapy unless the disease recurrence is histologically confirmed Surgery: No prior surgery (except biopsy) for recurrent brain tumor At least 3 months since prior surgery for primary brain tumor Other: No other concurrent anticancer agents No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2001-01; Primary Completion 2001-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin J. van Den Bent, MD, Study Chair — Daniel Den Hoed Cancer Center at Erasmus Medical Center
Locations (18):
- Kaiser Franz Josef Hospital, Vienna (Wien), Austria
- France (8):
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre de Lute Contre le Cancer,Georges-Francois Leclerc, Dijon
  - Centre Leon Berard, Lyon
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Centre Antoine Lacassagne, Nice
  - CHU Pitie-Salpetriere, Paris
  - Centre Eugene Marquis, Rennes
  - Institut Gustave Roussy, Villejuif
- University of Ioannina, Ioannina, Greece
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel
- Italy (2):
  - Azienda Ospedaliera di Padova, Padova (Padua)
  - Istituti Fisioterapici Ospitalieri - Roma, Rome
- Netherlands (2):
  - Rotterdam Cancer Institute, Rotterdam
  - Academisch Ziekenhuis Utrecht, Utrecht
- Instituto Portugues de Oncologia de Francisco Gentil, Lisbon, Portugal
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital - St. Gallen, Sankt Gallen